CLINICAL TRIAL: NCT06068075
Title: Liquid Biopsy in Ewing Sarcoma and Osteosarcoma as a Prognostic And Response Diagnostic: The LEOPARD Study
Brief Title: Liquid Biopsy in Ewing Sarcoma and Osteosarcoma as a Prognostic And Response Diagnostic: LEOPARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Alex's Lemonade Stand Foundation (Industry); Conquer Cancer Foundation (Other); Harvard University (Other); Sam Day Foundation (Unknown)
Responsible Party: Principal Investigator, David S Shulman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-138
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ewing Sarcoma; Ewing Sarcoma of Bone; Ewing Sarcoma of Soft Tissue; Peripheral Primitive Neuroectodermal Tumor; Peripheral Primitive Neuroectodermal Tumor of Bone; Peripheral Primitive Neuroectodermal Tumor of Soft Tissue; High-grade Osteosarcoma
Keywords: Ewing Sarcoma; Ewing Sarcoma of Bone; Ewing Sarcoma of Soft Tissue; Peripheral Primitive Neuroectodermal Tumor; Peripheral Primitive Neuroectodermal Tumor of Bone; Peripheral Primitive Neuroectodermal Tumor of Soft Tissue; High-grade osteosarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REG EWING or OSTEO: ctDNA EVALUATION (No Intervention): This study involves collection of blood samples at pre-specified time points as well as collection of information about this disease.
  For each timepoint, submit two tubes of blood (17 mL total or a little more than 3 teaspoons) per standard ctDNA workflow
- EWING ctDNA RETURN OF RESULTS (Experimental): This study involves collection of blood samples at pre-specified time points as well as collection of information about this disease.
  For each timepoint, submit two tubes of blood (17 mL total or a little more than 3 teaspoons) to a commercial testing laboratory called Foundation Medicine and one tube of blood (10 mL or 2 teaspoons) to standard ctDNA workflow
  Interventions: Other: FoundationOne Liquid CDx

INTERVENTIONS:
Other: FoundationOne Liquid CDx — a FoundationOne liquid biopsy test kit will be sent to the laboratory of the subject's treating center, in addition to the paired cell stabilizing tube from the primary center
  Other Names: Liquid Biopsy
  Arms: EWING ctDNA RETURN OF RESULTS

SUMMARY:
This is a prospective multicenter biomarker study evaluating the prognostic impact of ctDNA detection at diagnosis in patients with Ewing sarcoma or osteosarcoma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether ctDNA in the blood can provide information about the chances of Ewing sarcoma or osteosarcoma coming back after treatment. This research study is evaluating a new advanced laboratory test to detect small pieces of tumor genes in the peripheral blood known as circulating tumor DNA (ctDNA).

Part A : During this part of the research study (Part A) participants will be asked to provide blood samples at pre-defined times. These blood samples may help find specific genetic alterations commonly seen in Ewing sarcoma or osteosarcoma that may allow investigators to learn more about the uses of ctDNA. The results of the ctDNA analysis will not be returned to participants.

Approximately 90 patients will take part in this study across multiple centers.

Part B: This research study is evaluating new advanced laboratory tests to detect small pieces of tumor genes in the peripheral blood known as circulating tumor DNA (ctDNA). Part B of the research study, which focuses on ctDNA tests that can be returned to providers and patients with Ewing sarcoma. This part of the study will allow comparison of commercial ctDNA testing from Foundation Medicine to our research testing. It is expected that about 60 people with Ewing sarcoma will take part in Part B of this research study.

The sponsor of this protocol is Dana-Farber Cancer Institute and is providing funding for the study. Additional funding for this study is provided by the Conquer Cancer Foundation of the American Society of Clinical Oncology, Alex's Lemonade Stand Foundation, Boston Children's Hospital Office of Faculty Development, the Friends of Dana-Farber Cancer Institute, The Harvard Catalyst Program, and the Spada Pediatric Sarcoma Foundation

ELIGIBILITY:
Inclusion Criteria:

* For Part A, subjects must meet all of the following eligibility criteria.
* Age: ≥ 12 months of age at time of study enrollment to 50 years of age
* Diagnosis: Patients with histologic diagnosis (by institutional pathologist) of newly diagnosed, localized or regionally disseminated Ewing sarcoma or peripheral primitive neuroectodermal tumor (PNET) of bone or soft tissue or; Patients with histologic diagnosis (by institutional pathologist) of newly diagnosed, non-pelvic, localized or regionally disseminated high-grade osteosarcoma. NOTE: Staging will be assessed according to standard of care at the treating center.
* Prior Therapy:

  * Patients should have only previously had a biopsy, and not had prior attempt at tumor resection.
  * Not yet started chemotherapy or radiation therapy OR patient has started chemotherapy or radiation therapy, but an appropriate pre-treatment baseline sample was collected and processed for ctDNA under a local banking study in DFCI Pediatrics and is available to use for this study.
* Planned to receive chemotherapy as follows:

  -- VDC/IE as per COG protocols AEWS0031, AEWS1031 or AEWS1221 (for patients with Ewing sarcoma or PNET); or MAP as per COG protocol AOST0331 (for patients with osteosarcoma).
* For Part B subjects must meet all of the following eligibility criteria.
* Age: ≥ 12 months of age at time of study enrollment
* Diagnosis: Patients with histologic diagnosis (by institutional pathologist) of newly diagnosed Ewing sarcoma or peripheral primitive neuroectodermal tumor (PNET) of bone or soft tissue
* Prior Therapy:

  * Patients should have had only frontline therapy as per institutional standard, and maintenance therapy if given (no relapse therapy).
  * If frontline systemic therapy already completed (not including maintenance or metastatic site radiation), therapy completed within 6 months of enrollment to Part B.
  * Subjects must have a willing physician provider supporting their participation in Part B.
* For Part B, providers are eligible to receive the provider survey if they are listed as the primary provider for the patient at the study site.

Exclusion Criteria:

* For Part A, subjects must not meet any of the following exclusion criteria.
* Patients with distant metastatic disease.
* Patients with known Ewing-like sarcoma (e.g., BCOR-CCNB3 or CIC-DUX4 translocated small round cell sarcomas) are not eligible.
* Patients who are enrolled with an initial diagnosis of Ewing sarcoma and subsequently found to have Ewing-like sarcoma will be replaced. Samples obtained prior to removal from study will be analyzed and reported descriptively. Patients with Ewing-like tumors may continue to provide samples and clinical data until they meet off-study criteria per protocol.
* Patients weighing < 5 kg at time of diagnosis
* Patients with a second malignant neoplasm
* Patients without detectable tumor at the time of study enrollment (ie, complete tumor resection prior to study enrollment)
* Patients already receiving tumor-directed therapy at the time of study enrollment except when a pre-treatment baseline sample has already been obtained under a local banking study in DFCI Pediatrics that would be eligible for analysis under this study.
* Patients with osteosarcoma with a pelvic primary tumor site Pregnancy
* For Part B, subjects must not meet any of the following exclusion criteria.
* Patients with known Ewing-like sarcoma (e.g., BCOR-CCNB3 or CIC-DUX4 translocated small round cell sarcomas) are not eligible.
* Samples obtained prior to removal from study will be analyzed and reported descriptively. Patients with Ewing-like tumors may continue to provide samples and clinical data until they meet off-study criteria per protocol
* Patients weighing < 5 kg at time of enrollment
* Patients diagnosed with relapsed disease and/or having started therapy directed at disease relapse
* Pregnancy
* Resides outside of the United States
* For Part B, providers at non-study centers will not be eligible to receive the provider survey.

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 340 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival rate | 2 years
  Proportion of patient without an event by baseline detection of ctDNA

SECONDARY OUTCOMES:
Event-free survival rate | 2 years
  Proportion of patient without an event by ctDNA burden at baseline

CONTACTS AND LOCATIONS:
Overall Officials: David S Shulman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (15):
- United States (15):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital's and Clinics of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Lifespan / Rhode Island Hospital, Providence, Rhode Island
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah Childrens Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu